CLINICAL TRIAL: NCT05803629
Title: Characterizing Histiocytosis With 68Ga-FAPI PET/CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCHFAPIhistiocytosis
Record Dates: First submitted 2023-03-25; First posted 2023-04-07 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Histiocytosis
Keywords: histiocytosis; 68Ga-FAPI; PET/CT
MeSH Terms: conditions — Histiocytosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI ,PET/CT (Experimental): Inject 68Ga-FAPI and then perform PET/CT scan.
  Interventions: Diagnostic Test: 68Ga-FAPI; Diagnostic Test: 18F-FDG

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI — Intravenous injection of one dosage of 74-148 MBq(2-4 mCi) 68Ga-FAPI.
  Other Names: 68Ga-fibroblast activating protein inhibitors
Diagnostic Test: 18F-FDG — Intravenous injection of one dosage of 7.4MBq/kg(0.2mCi/kg) 18F-FDG. 18F-FDG PET/CT is performed within one week from 68Ga-FAPI PET/CT scan.

SUMMARY:
Histiocytic disorders are rare diseases that are characterized by tissue infiltration of histiocytes (dendritic cells) and other inflammatory white blood cells.68Ga-FAPI has been developed as a tumor-targeting agent as fibroblast activation protein is overexpressed in cancer-associated fibroblasts and it might be a pan-tumor PET agent.Recent discoveries have shown that inflammation and fibrosis secondary to mutated histiocytes, rather than a proliferative cell mechanism, result in manifestation of the disease.Thus, the investigators aim to carry out this prospective study to investigate the role of 68Ga-FAPI PET/CT in the diagnosis, therapy response assessment and follow-up of histiocytosis.

DETAILED DESCRIPTION:
Histiocytic disorders are rare diseases that are characterized by tissue infiltration of histiocytes (dendritic cells) and other inflammatory white blood cells. The archaic term "histiocyte" refers to large white blood cells resident in tissues and includes Langerhans cells, monocytes/macrophages, and dermal/interstitial dendritic cells. The Histiocytic Society classification divides histiocytic disorders into five categories, based on clinical, histologic, immunophenotypic, and molecular features. They are langerhans (L) group, cutaneous and mucocutaneous (C) group, Rosai-Dorfman disease (R) group, malignant histiocytosis (M) group and hemophagocytic lymphohistiocytosis (H) group. Langerhans cell histiocytosis is the most common histiocytic disorder. Less common types include Erdheim-Chester disease, Rosai-Dorfman disease, adult and juvenile xanthogranuloma. Diagnosis, which relies on a multidisciplinary approach, is challenging and often delayed because clinical findings are nonspecific and may mimic malignant processes at radiologic evaluation. Compared with conventional imaging, PET/CT allows detection of the increased metabolic activity in histiocytes and provides a comprehensive whole-body evaluation of their potential involvement with multiple organ systems and allows monitoring of therapeutic response. However, one drawback is that the uptake of FDG is nonspecific because histiocytic lesions may mimic neoplastic processes at PET/CT. And the physiological FDG metabolism in brain, liver and gastrointestinal tract, et al. hampers the detection rate of lesions located in these organs.68Ga-FAPI has been developed as a tumor-targeting agent as fibroblast activation protein is overexpressed in cancer-associated fibroblasts and it might be a pan-tumor PET agent. Although the pathogenesis of histiocytosis may be attributable to mutations in the oncogenic driver, recent discoveries have shown that inflammation and fibrosis secondary to mutated histiocytes, rather than a proliferative cell mechanism, result in manifestation of the disease. Considering 68Ga-FAPI revealing cancer-associated fibroblasts, the investigators aim to carry out this prospective study to investigate the role of 68Ga-FAPI PET/CT in the diagnosis, therapy response assessment and follow-up of histiocytosis.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed untreated histiocytosis patients
* 18F-FDG PET/CT within two weeks;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* known allergy against FAPI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 1 year
  Sensitivity and Specificity of 68Ga-FAPI PET/CT for histiocytosis in comparison with 18F-FDG PET/CT

SECONDARY OUTCOMES:
Metabolic parameters | through study completion, an average of 1 year
  Total Lesion Glycolysis (TLG) of histiocytosis lesions are measured on 68Ga-FAPI PET/CT.
FAPI expression and SUV | through study completion, an average of 1 year
  Correlation between FAPI expression and SUV in PET
Disease burden assessement | through study completion, an average of 1 year
  Correlation between Total Lesion Glycolysis (TLG) of histiocytosis lesions assessed on 68Ga-FAPI PET/CT and clinical parameters for histiocytosis
therapy response | through study completion, an average of 1 year
  Decrease of Total Lesion Glycolysis (TLG) on 68Ga-FAPI PET/CT after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yaping Luo, MD, Principal Investigator — Peking Union Medical College Hospital; Li Huo, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Department of Nuclear Medicine, Peking Union Medical College Hopital, Chinese Academy of Medical Science, Beijing, China